CLINICAL TRIAL: NCT06597799
Title: Phase 1, First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose, Multiple Ascending Dose, and Food-Effect Study to Assess Safety, Tolerability, PK and PD of MRT-6160 in Healthy Subjects
Brief Title: First-in-human Study of MRT-6160 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Monte Rosa Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRT-6160-001
Record Dates: First submitted 2024-08-02; First posted 2024-09-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: MRT-6160; MRT-6160-001; MRT; Monte Rosa Therapeutics; Healthy Volunteers; Single Ascending Dose; Multiple Ascending Dose; SAD; MAD

STUDY DESIGN:
Intervention Model Description: Sequential Ascending Doses, Multiple Ascending Doses
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single Ascending Dose (Experimental): Single Ascending Dose of either:
  MRT-6160 or matching placebo
  Interventions: Drug: MRT-6160; Drug: Placebo
- Multiple Ascending Dose (Experimental): Multiple Ascending Dose of either:
  MRT-6160 or matching placebo
  Interventions: Drug: MRT-6160; Drug: Placebo

INTERVENTIONS:
Drug: MRT-6160 — Orally administered tablets or capsules of MRT-6160
Drug: Placebo — Orally administered tablets or capsules of placebo

SUMMARY:
The principal aim of this study is to obtain safety and tolerability data when MRT-6160 is administered orally as single and multiple doses to healthy subjects. This information, together with the pharmacokinetic (PK) data, will help establish the doses and dosing regimen suitable for future studies in patients.

The study drug, MRT-6160, is experimental. This is the first study in which MRT-6160 will be given to humans.

Part 1: Subjects will receive a single oral dose of MRT-6160 or placebo on Day 1

Part 2: Subjects will receive multiple oral doses of MRT-6160 or placebo for 7 consecutive days

DETAILED DESCRIPTION:
Detailed Description:

The purpose of this study is to:

Learn about the safety and tolerability of single and multiple ascending oral doses of MRT-6160 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or females 19-65 years of age
* Non smoker who has not used nicotine and tobacco containing products for at least 3 months prior to start of study
* Able to swallow oral medications
* Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease that will interfere with adherence to study protocol
* Underwent surgical intervention or an operation within 4 weeks prior to start of study
* Has active TB, latent TB, a history of TB, or had close contact with a person with active TB within 8 weeks prior to the first dosing
* Female subject with a positive pregnancy test or who is lactating
* Positive urine drug or alcohol screen results
* Positive COVID-19 results indicating recent or current COVID-19
* Positive results for human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus or history of resolved hepatitis
* Participation in another clinical study within 30 days or within 5 half-lives (if known) prior to start of study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single ascending doses of MRT-6160 in healthy adult subjects | 6 weeks
  Frequency of adverse events as assessed by the National Cancer Institute - Common Terminology Criteria for Adverse Events Version 5.0
To evaluate the safety and tolerability of multiple ascending doses of MRT-6160 in healthy adult subjects | 7.5 weeks
  Frequency of adverse events as assessed by the National Cancer Institute - Common Terminology Criteria for Adverse Events Version 5.0

SECONDARY OUTCOMES:
To evaluate the effects of single dose or multiple doses of MRT-6160 on the heart rate (HR)-corrected QT (QTc) interval by assessing the concentration QT (C-QT) relationship using exposure-response modelling in healthy adult subjects. | 6 - 8 weeks
To characterize the PK profile of MRT-6160 in plasma after single or multiple doses of MRT-6160 in healthy adult subjects, with and without high fat/high calorie meal | 6 - 8 weeks
  Peak plasma Concentration (Cmax)
To characterize the PK profile of MRT-6160 in plasma after single or multiple doses of MRT-6160 in healthy adult subjects, with and without high fat/high calorie meal | 6 - 8 weeks
  Area under the plasma concentration versus time (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: CRO, Principal Investigator — Celerion
Locations (2):
- United States (2):
  - Celerion, Inc., Tempe, Arizona
  - Celerion, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: No